CLINICAL TRIAL: NCT02408289
Title: A Pilot Randomized Human Trial on The Effects of Cocoa on Appetite.
Brief Title: The Randomized Controlled Cocoa-Appetite Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooklyn College of the City University of New York (Other)
Responsible Party: Principal Investigator, James Greenberg, Associate Professor, Department of Health & Nutrition Sciences,, Brooklyn College of the City University of New York
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: PSC-CUNY 66522-0044
Record Dates: First submitted 2015-04-02; First posted 2015-04-03 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Catechin; Proanthocyanidins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lo-Flav (Placebo Comparator): Low-flavonoid cocoa powder with 0 mg of procyanidins and 0 mg epicatechin per kg of body weight will be consumed as a beverage
  Interventions: Dietary Supplement: Lo-Flav
- Hi-Flav (Active Comparator): Cocoa powder with 3.8 mg procyanidins per kg of body weight and 0.6 mg Epicatechin per kg of body weight will be consumed as a beverage.
  Interventions: Dietary Supplement: Hi-Flav
- Epicatechin (Active Comparator): Low-flavonoid cocoa powder plus 1 mg epicatechin per kg of body weight will be consumed as a beverage.
  Interventions: Dietary Supplement: Epicatechin
- Procyanidins (Active Comparator): Low-flavonoid cocoa powder plus 3.7 mg procyanidins per kg of body weight will be consumed as a beverage.
  Interventions: Dietary Supplement: Procyanidins

INTERVENTIONS:
Dietary Supplement: Lo-Flav — low-flavonoid cocoa powder with 0 mg of procyanidins and 0 mg epicatechin per kg of body weight will be consumed as a beverage.
  Arms: Lo-Flav
Dietary Supplement: Hi-Flav — High-flavonoid cocoa powder with 3.8 mg procyanidins per kg of body weight and 0.6 mg Epicatechin per kg of body weight will be consumed as a beverage.
  Arms: Hi-Flav
Dietary Supplement: Epicatechin — Low-flavonoid cocoa powder plus 1 mg epicatechin per kg of body weight will be consumed as a beverage
  Arms: Epicatechin
Dietary Supplement: Procyanidins — Low-flavonoid cocoa powder plus 3.7 mg procyanidins per kg of body weight will be consumed as a beverage.
  Arms: Procyanidins

SUMMARY:
The purpose of this study is to determine whether high-flavonoid cocoa can decrease appetite in humans. In addition the study is designed to test epicatechin, a compound found in cocoa and procyanidins, a class of compounds found in cocoa, for their ability to decrease appetite in humans.

DETAILED DESCRIPTION:
The study is a four-way randomized double-blinded crossover trial with randomization balanced for beverage and lab visit order.

ELIGIBILITY:
Inclusion Criteria:

* stable-weight, as indicated by weight gain or loss of <2% in the past 6 months;
* engaging in only mild exercise< twice a week;
* moderate alcohol users, <2 drinks/day;
* willing to eat pizza.
* mentally and physically healthy.

Exclusion Criteria:

* smokers regular;
* frequent drinkers of coffee, tea or cola sodas, >daily;
* underweight or obese (BMI: <18.5 or >30 Kg/m2);
* allergies to chocolate, cocoa, green tea, coffee or pizza;
* using medication;
* interested in registering in the future for the course Health & Nutrition Sciences 2140, Introduction to the U.S. Health Care System, that is often taught by the PI of the proposed study

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Appetite as assessed by amount of pizza eaten. | Two and a half hours
  Amount of pizza eaten to be assessed two and one half hours after ingestion of the beverage.

SECONDARY OUTCOMES:
Appetite as assessed by a Visual Analog Scale | Two and one half hours
  Visual Analog Scale assessments to be conducted during the two and one half hours after ingestion of the beverage.

CONTACTS AND LOCATIONS:
Overall Officials: James Greenberg, Ph.D, Principal Investigator — Department of Health & Nutritional Sciences, Brooklyn College of the City University of New York
Locations (1):
- Brooklyn College of the City University of New York, Brooklyn, New York, United States

REFERENCES:
- [Derived] Greenberg JA, O'Donnell R, Shurpin M, Kordunova D. Epicatechin, procyanidins, cocoa, and appetite: a randomized controlled trial. Am J Clin Nutr. 2016 Sep;104(3):613-9. doi: 10.3945/ajcn.115.129783. Epub 2016 Aug 10. PMID 27510533